CLINICAL TRIAL: NCT00745576
Title: An Open-label, Nonrandomized Study to Evaluate the Potential Pharmacokinetic Interaction Between Multiple Doses of Verapamil Immediate Release (IR) and a Single Dose of SAM-531 When Co-administered Orally to Healthy Young Adult Subjects
Brief Title: Study Evaluating The Potential Interaction Between Verapamil Immediate Release And SAM-531 When Co-Administered
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3193A1-1112
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2010-02-08 (Estimated); Status verified 2010-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SAM-531

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SAM-531

INTERVENTIONS:
Drug: SAM-531

SUMMARY:
The purpose of this study is to evaluate the effects of multiple doses of verapamil on the plasma concentration of a single dose of SAM-531 in healthy young adult subjects and to assess the safety and tolerability of co-administration of SAM-531 and verapamil.

ELIGIBILITY:
Inclusion criteria :

1. Body mass index in the range of 18 to 30 kg/m2 and body weight greater than 50 kg.
2. Healthy as determined by the investigator on the basis of medical history, physical examination findings, clinical laboratory test results, vital sign measurements, and digital 12-lead ECG readings.

Exclusion criteria :

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any significant cardiovascular, hepatic, renal, respiratory, gastrointestinal (GI), endocrine, immunologic, dermatologic, hematologic, neurologic, or psychiatric disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2008-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
blood samples | 7 weeks

SECONDARY OUTCOMES:
Safety based on supine vital signs evaluations, 12-lead ECGs and routine lab tests | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Gières, France